CLINICAL TRIAL: NCT02745899
Title: The Effect of Cow-milk Consumption on Respiratory Symptoms and Pulmonary Functions in Asthmatic and Non-asthmatic Children
Brief Title: The Effect of Cow Milk Consumption on Respiratory Symptoms and Pulmonary Functions in Asthmatic and Non Asthmatic Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: TASMC-16-KA-0070-16-TLV-CTIL
Record Dates: First submitted 2016-02-07; First posted 2016-04-20 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Asthma
Keywords: asthma; cow milk; pulmonary function testing; children; mucus
MeSH Terms: conditions — Asthma | interventions — Milk; Soy Milk

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Soy milk substitute Healthy (Active Comparator): Healthy children aged 6-18 will drink 240 ml of soy milk substitute.
  Interventions: Dietary Supplement: Soy milk
- Soy milk substitute Asthma (Active Comparator): Asthmatic children aged 6-18 will drink 240 ml of soy milk substitute.
  Interventions: Dietary Supplement: Soy milk
- Cow milk Healthy (Experimental): Healthy children aged 6-18 will drink 240 ml of cow milk.
  Interventions: Dietary Supplement: Cow milk
- Cow milk Asthma (Experimental): Asthmatic children aged 6-18 will drink 240 ml of cow milk.
  Interventions: Dietary Supplement: Cow milk

INTERVENTIONS:
Dietary Supplement: Cow milk — Ingestion of 240 ml cow milk
  Arms: Cow milk Asthma; Cow milk Healthy
Dietary Supplement: Soy milk — Ingestion of 240 ml soy milk
  Arms: Soy milk substitute Asthma; Soy milk substitute Healthy

SUMMARY:
the investigators hypothesis is that milk consumption, either in the acute phase and through prolonged exposure, does not cause or increase respiratory symptoms or airway inflammation. the investigators aim to objectively prove this by examining respiratory symptoms and signs and objectively measuring parameters of airway inflammation and hyper responsiveness after consumption of cow milk or soy milk substitute.

DETAILED DESCRIPTION:
In this prospective single blinded placebo controlled trial, acute milk consumption will be evaluated. 50 asthmatic and 50 healthy children aged 6-18 will drink 240 ml of cow milk or soy milk substitute. Respiratory symptoms by questionnaire and physical examination will be evaluated. Airway response and inflammation will be assessed by fraction of exhaled Nitric Oxide (FENO) and spirometry before and after the exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* Asthmatic children

Exclusion Criteria:

* Known allergy to cow milk
* Children had upper / lower respiratory disease in two weeks prior the study.
* Children who had been treated in systemic steroids in the month prior the study.
* Intolerant children to cow milk.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Cough and mucus production according to patient's report and physical examination | Baseline
  subjective report by the parents including: appearance of cough, rhinitis and objective physical examinations signs including: wheezing, rales, cough- yes or no
Cough and mucus production according to patient's report and physical examination | 30 minutes after the intervention
  subjective report by the parents including: appearance of cough, rhinitis and objective physical examinations signs including: wheezing, rales, cough- yes or no
Cough and mucus production according to patient's report and physical examination | 60 minutes after the intervention
  subjective report by the parents including: appearance of cough, rhinitis and objective physical examinations signs including: wheezing, rales, cough- yes or no
Cough and mucus production according to patient's report and physical examination | 90 minutes after the intervention
  subjective report by the parents including: appearance of cough, rhinitis and objective physical examinations signs including: wheezing, rales, cough- yes or no
Cough and mucus production according to patient's report and physical examination | 120 minutes after the intervention
  subjective report by the parents including: appearance of cough, rhinitis and objective physical examinations signs including: wheezing, rales, cough- yes or no

SECONDARY OUTCOMES:
Fraction of exhaled Nitric Oxide (FeNO) | Baseline
  single breath method: This test measures the concentration of NO in the exhaled air. In this method the patient takes a deep breath from the filter device and exhales the air at a constant rate of 50 mL / min for 12 seconds. The results of each test will be the average value of three tests.
  General measurement: overall system to be measured FENO device Denox 88 (ECO Medics AG, Switzerland), and nitric oxide 88 CLD analyzer which was approved for use by the FDA's medical device approval if the Ministry of Health. The values are in parts per billion (Ppb).
  children aged 5-6 years are able to perform this test.
  FENO values:
  Low FENO: 0-5 ppb in Children Normal FENO: 5-20 ppb in children Mild elevated FENO:20-30 ppb in children High FENO: 30-70 ppb in Children Severe FENO: >70 ppb in Children
Fraction of exhaled Nitric Oxide (FeNO) | 30 minutes after the intervention
  single breath method: This test measures the concentration of NO in the exhaled air. In this method the patient takes a deep breath from the filter device and exhales the air at a constant rate of 50 mL / min for 12 seconds. The results of each test will be the average value of three tests.
  General measurement: overall system to be measured FENO device Denox 88 (ECO Medics AG, Switzerland), and nitric oxide 88 CLD analyzer which was approved for use by the FDA's medical device approval if the Ministry of Health. The values are in parts per billion (Ppb).
  children aged 5-6 years are able to perform this test.
  FENO values:
  Low FENO: 0-5 ppb in Children Normal FENO: 5-20 ppb in children Mild elevated FENO:20-30 ppb in children High FENO: 30-70 ppb in Children Severe FENO: >70 ppb in Children
Fraction of exhaled Nitric Oxide (FeNO) | 60 minutes after the intervention
  single breath method: This test measures the concentration of NO in the exhaled air. In this method the patient takes a deep breath from the filter device and exhales the air at a constant rate of 50 mL / min for 12 seconds. The results of each test will be the average value of three tests.
  General measurement: overall system to be measured FENO device Denox 88 (ECO Medics AG, Switzerland), and nitric oxide 88 CLD analyzer which was approved for use by the FDA's medical device approval if the Ministry of Health. The values are in parts per billion (Ppb).
  children aged 5-6 years are able to perform this test.
  FENO values:
  Low FENO: 0-5 ppb in Children Normal FENO: 5-20 ppb in children Mild elevated FENO:20-30 ppb in children High FENO: 30-70 ppb in Children Severe FENO: >70 ppb in Children
Fraction of exhaled Nitric Oxide (FeNO) | 90 minutes after the intervention
  single breath method: This test measures the concentration of NO in the exhaled air. In this method the patient takes a deep breath from the filter device and exhales the air at a constant rate of 50 mL / min for 12 seconds. The results of each test will be the average value of three tests.
  General measurement: overall system to be measured FENO device Denox 88 (ECO Medics AG, Switzerland), and nitric oxide 88 CLD analyzer which was approved for use by the FDA's medical device approval if the Ministry of Health. The values are in parts per billion (Ppb).
  children aged 5-6 years are able to perform this test.
  FENO values:
  Low FENO: 0-5 ppb in Children Normal FENO: 5-20 ppb in children Mild elevated FENO:20-30 ppb in children High FENO: 30-70 ppb in Children Severe FENO: >70 ppb in Children
Fraction of exhaled Nitric Oxide (FeNO) | 120 minutes after the intervention
  single breath method: This test measures the concentration of NO in the exhaled air. In this method the patient takes a deep breath from the filter device and exhales the air at a constant rate of 50 mL / min for 12 seconds. The results of each test will be the average value of three tests.
  General measurement: overall system to be measured FENO device Denox 88 (ECO Medics AG, Switzerland), and nitric oxide 88 CLD analyzer which was approved for use by the FDA's medical device approval if the Ministry of Health. The values are in parts per billion (Ppb).
  children aged 5-6 years are able to perform this test.
  FENO values:
  Low FENO: 0-5 ppb in Children Normal FENO: 5-20 ppb in children Mild elevated FENO:20-30 ppb in children High FENO: 30-70 ppb in Children Severe FENO: >70 ppb in Children
Spirometry - Forced expiratory flow 1 sec | Baseline
  This test measures how much air is moved in and out of the lungs and how fast the air moves. the patient will be asked to take in a deep breath and to blow the air out into a filter that is connected to a computer. computer measures how much and how fast the air is blown out. Each test will be performed three times and the average value choice.Forced expiratory flow 1 sec (percent of predicted value) is the value that will be compared before and after the intervention.
Spirometry - Forced expiratory flow 1 sec | 30 minutes after the intervention
  This test measures how much air is moved in and out of the lungs and how fast the air moves. the patient will be asked to take in a deep breath and to blow the air out into a filter that is connected to a computer. computer measures how much and how fast the air is blown out. Each test will be performed three times and the average value choice.Forced expiratory flow 1 sec (percent of predicted value) is the value that will be compared before and after the intervention.
Spirometry - Forced expiratory flow 1 sec | 60 minutes after the intervention
  This test measures how much air is moved in and out of the lungs and how fast the air moves. the patient will be asked to take in a deep breath and to blow the air out into a filter that is connected to a computer. computer measures how much and how fast the air is blown out. Each test will be performed three times and the average value choice.Forced expiratory flow 1 sec (percent of predicted value) is the value that will be compared before and after the intervention.
Spirometry - Forced expiratory flow 1 sec | 90 minutes after the intervention
  This test measures how much air is moved in and out of the lungs and how fast the air moves. the patient will be asked to take in a deep breath and to blow the air out into a filter that is connected to a computer. computer measures how much and how fast the air is blown out. Each test will be performed three times and the average value choice.Forced expiratory flow 1 sec (percent of predicted value) is the value that will be compared before and after the intervention.
Spirometry - Forced expiratory flow 1 sec | 120 minutes after the intervention
  This test measures how much air is moved in and out of the lungs and how fast the air moves. the patient will be asked to take in a deep breath and to blow the air out into a filter that is connected to a computer. computer measures how much and how fast the air is blown out. Each test will be performed three times and the average value choice.Forced expiratory flow 1 sec (percent of predicted value) is the value that will be compared before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Keren Armoni Domany, Doctor, Principal Investigator — Department of Pediatric Pulmonology, Critical Care and Sleep Medicine Dana-Dwek Children's Hospital, Tel Aviv Sourasky Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koren Y, Armoni Domany K, Gut G, Hadanny A, Benor S, Tavor O, Sivan Y. Respiratory effects of acute milk consumption among asthmatic and non-asthmatic children: a randomized controlled study. BMC Pediatr. 2020 Sep 12;20(1):433. doi: 10.1186/s12887-020-02319-y. PMID 32919454